CLINICAL TRIAL: NCT02610361
Title: A Phase 1A/1B, Open-Label, Multiple-Dose, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics and Preliminary Antitumor Activities of the B RAF Inhibitor BGB 283 in Subjects With Solid Tumors
Brief Title: Study of the Safety and Pharmacokinetics of BGB-283 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-283-AU-001; ACTRN12614001176651 (Registry Identifier: The Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — BGB-283

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BGB-283 (Experimental)
  Interventions: Drug: BGB-283

INTERVENTIONS:
Drug: BGB-283 — In the dose escalation part(phase 1a): the dose levels will be escalated following a modified 3+3 dose escalation scheme.
  In dose expansion phase(Phase 1b): Patients will be assigned to different groups based on their tumor types

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetic profile and treatment effect of a new drug known as BGB-283 in patients with solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent prior to enrollment.
2. Male or female and at least 18 years of age.
3. A life expectancy of at least 12 weeks.
4. Histologically or cytologically confirmed advanced or metastatic solid tumor for which no effective standard therapy is available.
5. One of B-RAF, N-RAS, or K-RAS mutation positive solid tumor.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. Able to swallow and retain oral medication.
8. Adequate bone marrow, liver, and renal function:

   * Hemoglobin > 9 g/dL
   * Absolute neutrophil count ≥ 1000/mm^3
   * Platelets ≥ 100,000/mm^3
   * Total bilirubin ≤1.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with known liver metastasis)
   * Creatinine clearance ≥ 45 mL/min (calculated by the Cockcroft Gault formula).
9. Female subjects are eligible to enter and participate in the study if they are of:

   a) Non childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who

   i) Has had a hysterectomy,

   ii) Has had a bilateral oophorectomy (ovariectomy),

   iii) Has had a bilateral tubal ligation, or

   iv) Is post menopausal (total cessation of menses for ≥ 1 year).

   b) Childbearing potential, has a negative serum pregnancy test at screening (within 7 days of the first investigational product administration), and uses adequate contraception before study entry and throughout the study until 28 days after the last investigational product administration. Adequate contraception, when used consistently and in accordance with both the product label and the instructions of the physician, are defined as follows:

   i) Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.

   ii) Any intrauterine device with a documented failure rate of less than 1% per year.

   iii) Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.
10. Subjects with treated brain metastasis are eligible to enter and participate in the study if they are neurologically stable.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Subjects receiving cancer therapy (chemotherapy or other systemic anti cancer therapies, immunotherapy, radiation therapy, or surgery) at the time of enrollment.
3. Any major surgery within 28 days prior to enrollment.
4. Any radiotherapy within 14 days prior to enrollment, providing the subject has recovered from all toxicities to NCI-CTCAE ≤ Grade 1.
5. Use of any investigational anti cancer drug within 28 days before the first investigational product administration.
6. Unresolved toxicity > Grade 1 (according to NCI-CTCAE, Version 4.03) from previous anti cancer therapy, unless agreed by the sponsor.
7. History or presence of gastrointestinal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
8. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug or to any component of BGB-283. (To date there are no known Food and Drug Administration [FDA] approved drugs chemically related to BGB-283).
9. Untreated leptomeningeal or brain metastasis. Subjects with previously treated brain metastasis that are asymptomatic, off steroids for longer than 28 days are permitted.
10. Any unstable, pre-existing major medical condition that in the opinion of the Investigator contra indicates the use of an investigational product, including active infection, known human immunodeficiency virus (HIV) positive subjects, or known Hepatitis B or C.
11. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
12. As a result of the medical interview, physical examination or screening investigations, the investigator considers the subject unfit for study.
13. Is on medication listed in the protocol or requires any of these medications during treatment with BGB-283.
14. Candidates for curative therapy.
15. Unable or unwilling to comply with the required treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events in phase 1a | From first dose to within 28 days of last dose of BGB-283, within 1 years in average
Objective response rate based on RECIST Version 1.1 in subjects with selected tumor types in phase 1b | From the first administration of the investigational product to the end of the study treatment, within 1 year in average

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the time of the last measurable concentration (AUClast) in phase 1a | During first 2 weeks
Area under the plasma concentration-time curve from time 0 to infinity time in (AUC∞) in phase 1a | During first 2 weeks
Maximum plasma concentration (Cmax) in phase 1a | During first 2 weeks
Time to reach maximum plasma concentration (tmax) in phase 1a | During first 2 weeks
Terminal elimination half-life (t1/2) in phase 1a | During first 2 weeks
Tumor response in phase 1a | Every 6 weeks from first dose until the date of first documented progression or date of death from any cause, whichever came first, within 1 year in average
Number of participants with adverse events in phase 1b | From first dose to within 28 days of last dose of BGB-283, within 1 year in average
Progression-free survival (PFS) | The interval from study treatment initiation until the determination of disease progression or death, within 1 year in average

CONTACTS AND LOCATIONS:
Overall Officials: Jayesh Desai, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (19):
- Australia (15):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - North Coast Cancer Institute, Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Tasman Oncology Research Ltd, Southport Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Alfred Cancer Trials, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton Waikato
  - Wellington Regional Hospital (Ccdhb), Wellington

IPD SHARING:
Plan to Share IPD: Yes
Upon request, and subject to certain criteria, conditions, and exceptions, BeiGene will provide access to individual de-identified participant data from BeiGene-sponsored global interventional clinical studies conducted for medicines for indications that have been approved or in programmes that have been terminated. BeiGene will also consider requests for the protocol, data dictionary, and statistical analysis plan. Data requests can be submitted to medicalinformation@beigene.com.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Desai J, Gan H, Barrow C, Jameson M, Atkinson V, Haydon A, Millward M, Begbie S, Brown M, Markman B, Patterson W, Hill A, Horvath L, Nagrial A, Richardson G, Jackson C, Friedlander M, Parente P, Tran B, Wang L, Chen Y, Tang Z, Huang W, Wu J, Zeng D, Luo L, Solomon B. Phase I, Open-Label, Dose-Escalation/Dose-Expansion Study of Lifirafenib (BGB-283), an RAF Family Kinase Inhibitor, in Patients With Solid Tumors. J Clin Oncol. 2020 Jul 1;38(19):2140-2150. doi: 10.1200/JCO.19.02654. Epub 2020 Mar 17. PMID 32182156